CLINICAL TRIAL: NCT03760432
Title: Clinical Trial of Laser Custom Corneal Collagen Cross-Linking in Keratoconus
Brief Title: Collagen Cross-linking in Keratoconus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, Peterson Professor of Ophthalmology & Professor of Biomedical Engineering, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6612-CXL; R01EY028755 (NIH)
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Keratoconus
Keywords: Keratoconus (KCN); Optical Coherence Tomography (OCT); Collagen Cross-linking (CXL)
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Surgery (Experimental): OCT-guided custom laser CXL
  Interventions: Procedure: Laser Custom Corneal Collagen Cross-Linking

INTERVENTIONS:
Procedure: Laser Custom Corneal Collagen Cross-Linking — Preoperative measurements from the OCT are used to assist the calculation in deciding the laser depth settings for smoothing the anterior corneal surface and removing any present opacities. The surgeon uses the OCT data to plan treatment parameters while preserving at least 360 microns of residual corneal stroma using a phototherapeutic keratectomy procedure. After the laser procedure, adjunctive MMC or saline solution will be applied to the cornea in accordance with the group to which the treated eye is randomized. The CXL procedure is then performed following the FDA-approved CXL regimen by Avedro, Inc.

SUMMARY:
Optical Coherence Tomography (OCT) devices are non-contact instruments that can measure the depth of scars, other causes of cloudiness of the cornea, and degree of corneal thinning in patients with keratoconus. Laser Custom Corneal Collagen Cross-linking (CXL) significantly decreases corneal aberrations and improves vision. This study will use OCT-guided setting for the lasers used in the corneal smoothing portion of the laser custom CXL procedure to assess the affect on visual outcomes.

DETAILED DESCRIPTION:
In the U.S., CXL and topography-guided laser ablation were approved independently, but not together. Another variation in technique involves the use of mitomycin-C (MMC), which is effective in reducing corneal haze after the laser surface ablation. Use of MMC during the laser custom CXL was associated with better outcomes, but in separate trials that could not be directly compared. This study will use OCT measurements to evaluate the magnitudes of direct and indirect laser actions after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of keratoconus
* Minimum corneal thickness of 410 microns

Exclusion Criteria:

* Inability to maintain fixation for OCT imaging
* Inability to commit to required study visits
* Inability to give informed consent
* Eyes with concurrent retinal diseases, glaucoma, or other eye conditions that may limit the visual outcome after surgery
* Mature cataracts if found to limit visual potential to worse than 20/40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in best spectacle-corrected visual acuity after laser custom CXL | 6 months after the CXL procedure
  The primary goal of the trial is to determine the extent of visual improvement after laser custom CXL compared to preoperative measurements. Vision will be checked at various time points, but the primary time point will be 6-months post-procedure.

SECONDARY OUTCOMES:
Determine CXL demarcation line depth | 1 month after the CXL procedure
  The study will use OCT imaging to measure the CXL demarcation line inside the entire optical zone. The demarcation line indicates the portion of corneal stroma being cross-linked. This helps determine to what extent the cornea is being strengthened.

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States